CLINICAL TRIAL: NCT05353218
Title: Efficacy of Ultrasound-Guided Intermediate Versus Deep Cervical Plexus Block for Carotid Endarterectomy: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Intermediate Versus Deep Cervical Plexus Block for Carotid Endarterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozlem Turhan, Specialist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/923
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia
Keywords: cervical plexus block; Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: Randomized, Prospective
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intermediate cervical plexus block (GI) (Active Comparator): Patients anesthetized with intermediate cervical plexus block.
  Interventions: Procedure: Intermediate cervical plexus block
- Group deep cervical plexus block (GD) (Active Comparator): Patients anesthetized with deep cervical plexus block.
  Interventions: Procedure: Deep cervical plexus block

INTERVENTIONS:
Procedure: Intermediate cervical plexus block — Intermediate cervical plexus block will be applied in transverse plane using posterior approach at C4.
  Arms: Group intermediate cervical plexus block (GI)
Procedure: Deep cervical plexus block — Deep cervical plexus block will be appliedin transverse plane using anterior approach at C2-3-4.
  Arms: Group deep cervical plexus block (GD)

SUMMARY:
Cervical plexus blocks are regional methods used in carotid endarterectomy. Cervical plexus blocks consist of three blocks: superficial, intermediate and deep. These three blocks can be used alone or combined. The aim of this study is to evaluate the effectiveness of ultrasound-guided intermediate and deed cervical plexus block in patients undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
Carotid endarterectomy is a surgical method used to treat occlusive lesions of the carotid. Regional anesthesia is preferred because it allows for consciousness control and neurological examination during the operation. Cervical plexus blocks are regional methods used in carotid endarterectomy. It is a regional technique in which the cervical spinal nerves (C2-C3-C4) are blocked with a local anesthetic agent from different regions. Cervical plexus blocks consist of three blocks: superficial, intermediate and deep, depending on the depth at which the local anesthetic agent is infiltrated. According to the preference of the clinician for the purpose of anesthesia, these three blocks can be used separately or combined. It is mentioned that all three blocks provide sufficient anesthesia for carotid endarterectomy surgery to be performed.

In the study, investigators planned to evaluate the effectiveness of ultrasound-guided intermediate and deep cervical plexus blocks in patients undergoing carotid endarterectomy by comparing the number of patients who need additional local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for carotid endarterectom y surgery.

Exclusion Criteria:

* Local infection
* Previous ipsilateral surgery
* Radiotherapy
* Conversion to general anesthesia
* Known bleeding disorders
* Known allergy of local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Number of patient needed supplemental local anesthetic | Intraoperative 2-3 hours
  If patients complain about pain above visual analog scale 3, 4ml 1% lidocaine is injected by surgeon.

SECONDARY OUTCOMES:
Amount of supplemental local anesthetic | Intraoperative 2-3 hours
  If patients complain about pain above visual analog scale 3, 4ml 1% lidocaine is injected by surgeon.
Duration of blocks' application | Up to 15 minutes
  time from the insertion of probe to the removal of needle from skin
Region where patient needs supplemental local anesthetic | Intraoperative 2-3 hours
  Region where supplemental lidocaine is injected by surgeon
Amount of remifentanil | Intraoperative 2-3 hours
  Amount of remifentanil (0.02mcg/kg/min) infused during surgery for sedation.
Pain assessment | Intraoperative 2-3 hours
  Pain assessment will be assessed using visual analog scale (VAS 0 to 10; 0: no pain, 10: the worst pain imaginable )
Complications | Up to 24 hours
  Hematoma, dysphagia, hoarseness, facial paralysis, Horner's syndrome, intravascular or intrathecal injection
Patient's satisfaction | Up to 24 hours
  Likert scale:1-5 (1: very dissatisfied, 5: very satisfied)
Surgeon's satisfaction | Up to 24 hours
  Likert scale:1-5 (1: very dissatisfied, 5: very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turhan O, Sivrikoz N, Canbolat N, Demirel EE, Altun D, Sungur Z. Ultrasound-guided intermediate versus deep cervical plexus block for carotid endarterectomy: a randomized controlled study. BMC Anesthesiol. 2025 Nov 21;25(1):581. doi: 10.1186/s12871-025-03460-w. PMID 41272478